CLINICAL TRIAL: NCT05381246
Title: The Effect of Reiki and Acupressure Applied After Percutaneous Coronary Intervention on Pain, Anxiety and Vital Signs During Femoral Catheter Extraction: A Randomized Controlled Trial.
Brief Title: The Effect of Reiki and Acupressure on Pain, Anxiety and Vital Signs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Abdullah Avcı, Nursing researcher, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MERSİN-AVCI-001
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Acupressure; Reiki; Pain; Anxiety; Vital Signs
MeSH Terms: conditions — Coronary Artery Disease; Pain; Anxiety Disorders | interventions — Acupressure; Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure group (Experimental): A total of 18 minutes of compression will be applied to each point for three minutes, as the Heart Meridian is at the 7th point (HT7), the Large Intestine Meridian is at the 4th point (LI4) and the pericardial meridian is at the 6th point (PC6).
  Interventions: Other: Acupressure
- Reiki group (Experimental): In the reiki group the crown chakra (top of the head), the forehead chakra (above the forehead), the throat chakra (above the throat), the heart chakra (the middle of the chest), the solar plexus (under the chest, above the navel), the sacral chakra (below the navel) and the root chakra (above the coccyx) will be applied to the region of the 7 chakra points on.In the reiki group, the reiki application time will take 21 minutes on average.
  Interventions: Other: Reiki
- Control group (No Intervention)

INTERVENTIONS:
Other: Acupressure — In the acupressure group, heart meridian 7th point (HT7), large intestine meridian 4th point, and pericardial meridian 6th point (PC6) will be applied. Tissue sensitivity will be reduced by heating and rubbing for about 20 seconds without direct pressure on the acupressure points, and the points will be ready for acupressure application. Subsequently, consecutive (breathing rhythm) compressions will be applied to the acupressure points determined by the researcher, without raising the finger, taking into account the pain threshold of the individual who is applied with the thumb, with 10 seconds of pressure for two seconds of relief Since the symmetry of the selected three different points will also be applied to the other extremity, a total of 18 minutes of compression will be applied to each point, provided that it is three minutes.
  Arms: Acupressure group
Other: Reiki — In the reiki group, the crown chakra (top of the head), the forehead chakra (above the forehead), the throat chakra (above the throat), the heart chakra (the middle of the chest), the solar plexus (under the chest, above the navel), the sacral chakra (below the navel) and the root chakra (above the coccyx) will be applied to the region of the 7 chakra points on.In the reiki group, the reiki application time will take 21 minutes on average.
  Arms: Reiki group

SUMMARY:
This research aims to determine the effects of reiki and acupressure applied after percutaneous coronary intervention on pain, anxiety and vital signs during femoral catheter extraction.

DETAILED DESCRIPTION:
In this study, 84 patients with percutaneous coronary intervention were assigned to the reiki, acupressure and control groups by block randomization method.In the acupressure group (n=28) the heart meridian 7th point (HT7) large intestine meridian 4th point (LI4) and pericardial meridian 6th point (PC6) will be applied to a total of three points.Depending on the preparation and compression time on each point, the session duration of each patient will be 18 minutes on average.In the reiki group (n=28) the crown chakra (top of the head), the forehead chakra (above the forehead), the throat chakra (above the throat), the heart chakra (the middle of the chest), the solar plexus (under the chest, above the navel), the sacral chakra (below the navel) and the root chakra (above the coccyx) will be applied to the region of the 7 chakra points on.In the reiki group, the reiki application time will take 21 minutes on average.Routine care will be applied to the control group (n=28).Pre-test data of patients in the acupressure, reiki and control groups will be collected 30 minutes before femoral catheter extraction after percutaneous coronary. Posttest data will be collected five minutes after femoral catheter extraction.

Data will be collected using the "Personal Information Form", "Visual Analog Scale", "State Anxiety Inventory" and "Vital Signs Evaluation Form".

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Percutaneous coronary intervention (PCI) for the first time,
* Previously planned PCI (elective patients),
* No additional procedure to percutaneous coronary intervention,
* Awake and conscious during percutaneous coronary intervention (not taking sedatives)
* A single sandbag is placed on the intervention area,
* Able to lie flat on his back (without respiratory distress),
* Hemodynamically stable (absence of chest pain and arrhythmia),
* No analgesic drug administered at least four hours before,
* No complications such as hematoma or bleeding in the operation area,
* No deformity or lesion in the areas where acupressure will be applied,
* No previous experience of acupressure and reiki application,
* Not diagnosed with anxiety disorder and not receiving medical treatment,
* Literate,
* Have sufficient communication skills and
* Those who signed the Informed Consent Form to participate

Exclusion Criteria:

* Emergency patients whose PCI was not planned beforehand,
* Bleeding, hematoma, etc. at the femoral intervention site during and after the procedure. developing complications,
* Any deformity, wound or lesion in the areas where acupressure will be applied,
* Coronary angiography only,
* Thrombocyte level less than 100,000 mg/dl,
* Those who did not sign the Informed Consent Form to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Pain evaluated using the Visual Analog Scale | 30 minutes
  The scale consists of a 10 cm ruler on which there is no pain on one end and excruciating pain on the other, on which the patient marks the pain. The distance between the point where the patient marked the pain and the pain-free interval is measured in cm and recorded.
Anxiety evaluated using the State Anxiety Inventory | 30 minutes
  The scale consists of 20 statements. The total score can range from 20 to 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Gün, Doctorate, Study Director — Mersin University

IPD SHARING:
Plan to Share IPD: No